CLINICAL TRIAL: NCT07053930
Title: To Compare the Mean Duration of Third Stage of Labour Between Intraumbilical and Intravenous Oxytocin.
Brief Title: Comparison of the Mean Duration of 3rd Stage of Labour Between Intraumbilical and Intravenous Oxytocin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRANAMJAVED
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraumbilical oxytocin group (Experimental): Patients were given 10 U of intraumbilical oxytocin, diluted in 10 mL of normal saline.
  Interventions: Drug: Intraumbilical oxytocin
- Intravenous oxytocin group (Experimental): Patients received 20 U of intravenous oxytocin diluted in 500 mL of normal saline.
  Interventions: Drug: Intravenous oxytocin

INTERVENTIONS:
Drug: Intraumbilical oxytocin — Patients were given 10 U of intraumbilical oxytocin, diluted in 10 mL of normal saline.
  Arms: Intraumbilical oxytocin group
Drug: Intravenous oxytocin — Patients received 20 U of intravenous oxytocin diluted in 500 mL of normal saline.
  Arms: Intravenous oxytocin group

SUMMARY:
There is always a debate for choosing the best method for management of the third stage of labour (TSL) in the general practice for reducing the duration of TSL. Although intravenous oxytocin is more extensively used in general practice for managing TSL than intraumbilical, it still needs to be properly investigated among local populations and in local settings.

DETAILED DESCRIPTION:
The findings of this study could identify the better route of oxytocin injection that could guide clinicians and health providers to opt for the better route in their routine practice for the management of TSL in order to reduce the morbidity and mortality of the patients, especially for developing countries like Pakistan, where most of the deliveries are conducted at peripheral or rural centers by a nurse, midwife, or a trained dai.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-40 years
* With spontaneous vaginal delivery
* Singleton pregnancy
* Gestational age >37 weeks
* Parity l-5
* Any gravidity

Exclusion Criteria:

* Females with intrauterine fetal death
* Malpresentation
* Multiple pregnancy
* Polyhydramnios
* Premature rupture of membranes
* Medical disorders and hypertensive disorders of pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Duration of the third stage labour | 30 minutes
  The duration of the third stage labour was measured from the completed delivery of the newborn until the completed delivery of the placenta.

CONTACTS AND LOCATIONS:
Overall Officials: Anam Javed, Principal Investigator — Sadiq Abbasi Hospital, Bahawalpur, Pakistan; Komal Iqbal, Principal Investigator — Sadiq Abbasi Hospital, Bahawalpur, Pakistan
Locations (1):
- Sadiq Abbasi Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.